CLINICAL TRIAL: NCT06488404
Title: Improving School Ethos Towards Mental Health Through Whole School Mental Health Interventions: Implementation Science Approach
Brief Title: Implementation Science to Improve School Ethos for Mental Health
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Schizophrenia Research Foundation (SCARF India), Chennai, India (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Other Study IDs: STUDY22120105; D43TW009114 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue
Keywords: Mental Health; School ethos; In depth interview
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to identify the challenges and opportunities existing within the school ethos in implementing evidence-based interventions to improve youth mental health and to identify the most appropriate implementation strategies for improving mental health among young people in schools at Chennai, a city in Southern part of India, a low- and middle- income country setting.

DETAILED DESCRIPTION:
The study team will approach the schools where the proposed study will take place and will obtain the needed permission to conduct the study in the school premises. Information about the study to all the potential participants will be disseminated through the school management. All the potential participants can approach the study team to learn more about the study and participate in the study. Potential participants approaching the study team will be explained in detail about the project and informed consent and /or assent will be obtained. The participants will be selected based on the proposed inclusion and exclusion criteria of the study.

After the recruitment of the participants, iIn-depth, semi-structured, individual interviews lasting approximately an hour will be conducted in either English or Tamil. This will be conducted by trained qualitative researchers. Interviews will be audiotaped and transcribed verbatim. A qualitative descriptive approach will guide all aspects of the qualitative methods we employ to derive a comprehensive description of participants' experiences that is both deep and meaningful. The IDI guide will be developed following an extensive literature search and discussions with experts in the field, for understanding the participants. The interviews will be conducted by two members of the research team. Face-to-face interviews or online interviews will be conducted after ensuring that the participant is comfortable, and all external disturbances will be taken care or minimized

ELIGIBILITY:
Inclusion Criteria:

* Students between 12-18 years of age
* Teachers 25-60 years of age
* Parents 25-60 years of age
* Management 25-60 years of age
* Mental health professionals 25-60 years of age
* School counsellors 25-60 years of age
* Education department - Government of Tamil Nadu 25-60 years of age
* Health department - Government of Tamil Nadu 25-60 years of age

Exclusion Criteria:

* Not willing to provide informed consent
* Can not speak either English or Tamil (native language)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All the interviews and the quantitative assessment will be conducted with the students, staff, parents, and management of the selected schools. Besides these, few interviews will be conducted with Government officials who are working with youth mental health and education, experts on school mental health and other relevant individuals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
School ethos | for six months
  Understanding the school ethos towards mental health prevailing in the schools from urban settings using in-depth interviews
Challenges and bariers | For six months
  Making a list of the challenges and opportunities in establishing and implementing a positive school ethos towards mental health in the schools using in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- Schizophrenia Research Foundation (SCARF India), Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.